CLINICAL TRIAL: NCT03116178
Title: Pleth Variability Index Based Intraoperative Fluid Management in Head and Neck Free Flap Reconstructive Surgeries
Brief Title: PVI Based Intraoperative Fluid Management in Head and Neck Free Flap Reconstructive Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, DR ITEE CHOWDHURY, Dr (senior consultant), Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RGCI ID:503/AN/ITC-02
Record Dates: First submitted 2016-11-11; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Free Tissue Flaps
Keywords: Fluid therapy; oximetry; thromboelastography; intraoperative/method; monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Active Comparator): Group B- intervention -Body weight guided Intraoperative fluid administered @ 6-8 ml/kg and blood loss replacement with colloid.
  hourly urine output if less than 0.5ml/hr 100-200ml bolus of plasmalyte was administered.
  Interventions: Other: Group B- Body weight guided intravenous fluid @6-8ml/kg
- Group G (Active Comparator): Group G- intervention - PVI( Masimo co oximeter) guided fluid therapy.
  Interventions: Other: Group G -PVI( Masimo co oximeter) guided fluid therapy

INTERVENTIONS:
Other: Group G -PVI( Masimo co oximeter) guided fluid therapy — goal directed fluid therapy maintaining pvi 4-11. when pvi<4 fluid rate is 50-60ml/hr and pvi>11 200ml colloid bolus transfusion till pvi value achieves normal range.
  In the control group crystalloid was administered @ 6-8 ml/kg and blood loss was replaced by colloids. Hourly urine output was measured and if less than 0.5ml/hr bolus crystalloid 100-200ml was administered
  Arms: Group G
Other: Group B- Body weight guided intravenous fluid @6-8ml/kg — Intravenous fluid @6-8ml.kg and blood loss replacement with colloids maintaining urine output of 0.5ml/kg
  Arms: Group B

SUMMARY:
Intraoperative fluid given according to BMI in group B and according to pulse oximeter- derived pleth variability index(MASIMO RAINBOW PULSE CO OXIMETRY) in group G. Comparison of haemodynamics, urine output,blood lactate levels, blood sugar, flap sugar and coagulation profile between the two groups.

DETAILED DESCRIPTION:
A sample size of 80 taken and computer generated random allocation done to divide the patients in two groups(40 each). Head and neck onco surgery patients undergoing resection and reconstruction with radial artery free flap and antero lateral thigh free flap of duration 4-6 hours taken for surgery.

Group B to receive intravenous fluid according to body weight stating at the rate 6-8 ml/kg/hr.

Group G to receive intravenous fluid according to Pleth variability index value(4-11).Blood loss up to 10% replacement by colloids.

Comparison of following parameters:

Demography, haemodynamics,urine output .blood lactate, ph, oxygenation index ,thromboelastography (TEG), blood sugar, flap sugar .

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing radial and anterolateral free flap

Exclusion Criteria:

* Duration of surgery > 6hrs
* BMI > 30
* Patients on anti platelet drugs
* Patient refusal

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in TEG waveform tracing as obtained from TEG 5000 Hemostasis analyser system | six months
  The investigators hypothesize that the patients in group G receiving PVI (pleth variability index) guided fluid therapy will have normal TEG parameter (R,K, ALPHA, MA and LY30) values and the patients in group B may have abnormal TEG parameter values.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Background] Yu Y, Dong J, Xu Z, Shen H, Zheng J. Pleth variability index-directed fluid management in abdominal surgery under combined general and epidural anesthesia. J Clin Monit Comput. 2015 Feb;29(1):47-52. doi: 10.1007/s10877-014-9567-5. Epub 2014 Feb 21. PMID 24557584